CLINICAL TRIAL: NCT02567266
Title: Community Study of Outcome Monitoring for Emotional Disorders in Teens
Acronym: COMET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: University of Connecticut (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Amanda Jensen-Doss, Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20150187; R01MH106536 (NIH); R01MH064089 (NIH)
Record Dates: First submitted 2015-10-01; First posted 2015-10-02 (Estimated); Results first posted 2021-08-18 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Unified Protocol for Adolescents (UP-A) (Experimental): Participants will be treated with the Unified Protocol for the Treatment of Emotional Disorders in Adolescence. Their clinicians will also receive feedback using the Youth Outcomes Questionnaire feedback system.
  Interventions: Behavioral: Unified Protocol for Adolescents (UP-A); Behavioral: Youth Outcomes Questionnaire
- Treatment as Usual Plus (TAU+) (Experimental): Participants will be treated by clinicians who receive feedback using the Youth Outcomes Questionnaire, but who otherwise use Treatment as Usual
  Interventions: Behavioral: Youth Outcomes Questionnaire; Behavioral: Treatment as Usual
- Treatment as Usual (TAU) (Active Comparator): Participants will receive Treatment as Usual provided at the study clinics.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Unified Protocol for Adolescents (UP-A) — The UP-A is an emotion-focused, transdiagnostic approach for adolescents (ages 12-18) with a primary emotional disorder. It is a developmental adaptation of the Unified Protocol, a transdiagnostic treatment for adults with emotional disorders. Clinicians present all skills in the context of the emotions most salient to presenting concerns and adolescent/caregiver conceptualizations of treatment needs, thereby personalizing treatment. The UP-A is delivered in 8-21 weekly sessions, with clinician flexibility regarding the sequencing and depth with which various sections are presented to clients and caregivers, as well as the emotions targeted during the course of the intervention.
  Arms: Unified Protocol for Adolescents (UP-A)
Behavioral: Youth Outcomes Questionnaire — The YOQ consists of parent- and youth-report measures of symptoms and alliance administered weekly on a tablet computer. The YOQ online system then generates reports to provide clinicians with systematic feedback about client progress, flagging "critical items" that have been endorsed (e.g., suicidality, hallucinations), presenting graphs of ratings over time, and providing empirically-derived "alerts" when clients are failing to progress or showing deterioration. Clinicians will be trained to use this feedback to modify treatment as needed, share it with families as appropriate, and use it to enhance use of supervision.
  Arms: Treatment as Usual Plus (TAU+); Unified Protocol for Adolescents (UP-A)
Behavioral: Treatment as Usual — Clinicians assigned to the TAU condition will be instructed to use whatever treatment methods and outcome monitoring strategies they typically use with adolescents with internalizing disorders.
  Arms: Treatment as Usual (TAU); Treatment as Usual Plus (TAU+)

SUMMARY:
This study is being done to compare three types of talk therapies for youth who struggle with emotional and behavioral problems (e.g., anxiety, sadness, worries) in Community Mental Health Clinics in Connecticut (CT) and Florida (FL).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adolescents between the ages of 12-18 years at the time of enrollment with clinically significant symptoms of anxiety or depression at baseline. Evidence of clinically significant symptoms will be defined as a Clinical Severity Rating (CSR) greater than or equal to 4 on any DSM-5 defined anxiety disorder (e.g., generalized anxiety disorder, social phobia, selective mutism, separation anxiety disorder) or depressive disorder (e.g., major depressive disorder, persistent depressive disorder), or an adjustment disorder with depressed mood, anxiety, or mixed anxiety and depressed mood.
2. The adolescent is determined by the community mental health center to be eligible for outpatient psychosocial services at the clinic and determined by the study IE to be appropriate for outpatient psychosocial intervention (e.g., no major cognitive impairment or active suicidality) based on clinical interview.
3. The adolescent lives (for at least 50% time) with legal guardian and this guardian is willing to attend treatment sessions and participate in study assessments (every effort will be made to encourage the same caregiver to participate in all assessments).
4. Adolescent and parent/guardian are able to complete all study procedures in English or Spanish.

Exclusion Criteria:

1. Adolescents will be excluded if they are receiving concurrent psychotherapy, family therapy or similar psychosocial interventions.
2. Consistent with the prior RCT of the UP-A, the use of psychopharmacologic treatments for anxiety or depression is allowable; but the adolescent must be on a stable dosage for 2 months for SSRI or 1 month for benzodiazepine prior to consenting to the study. The type, dosage and frequency of medication will be monitored at all major study assessment points, but subsequent changes will not incur exclusion from the investigation. Adolescents on stable doses of a stimulant for ADHD for at least one month or on a SNRI (e.g., Strattera) for ADHD for at least two months can also be included.
3. Adolescents who are currently suicidal or who have engaged in suicidal behaviors within the past 6 months will be excluded and referred for appropriate clinical intervention.
4. Adolescents with a current substance abuse disorder as determined using the ADIS-5-C/P, will be excluded.
5. Consistent with prior trials of the UP-A, youth with primary conditions not specified for exclusion (e.g., eating disorders, schizophrenia) will be screened. As long as study staff concur that an emotional disorder treatment focus is appropriate, these youth will be included.
6. Adolescents with a reported history of intellectual disability or for whom there is substantial evidence (e.g., multiple learning disorders, extensive school-based accommodations for learning) that the cognitive level of the UP-A would make it inappropriate as an individual therapy modality, as determined via Family Background Questionnaire and/or based on PI judgement, will be excluded.
7. Given additional complexities obtaining informed consent, adolescents who are currently placed in the foster care system will be excluded.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 196 (Actual)
Dates: Start 2016-01; Primary Completion 2020-07-30 (Actual); Study Completion 2020-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Golda Ginsburg, Ph.D., Principal Investigator — University of Connecticut; Amanda Jensen-Doss, Ph.D., Principal Investigator — University of Miami; Jill Ehrenreich-May, Ph.D., Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - University of Connecticut Health Center, West Hartford, Connecticut
  - University of Miami, Coral Gables, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ehrenreich-May J, Jensen-Doss A, Milgram L, Rosenfield D, Shaw AM, LoCurto J, Nanda Robinson M, Caron EB, Lee P, Ginsburg GS. A randomized controlled effectiveness trial of transdiagnostic treatment and measurement-based care for adolescents with emotional disorders in community clinics. J Consult Clin Psychol. 2025 Mar;93(3):144-160. doi: 10.1037/ccp0000947. PMID 40014505

RESULTS

PARTICIPANT FLOW:
Groups:
- Unified Protocol for Adolescents (UP-A): Participants will be treated with the Unified Protocol for the Treatment of Emotional Disorders in Adolescence (UP-A). Their clinicians will also receive feedback using the Youth Outcomes Questionnaire feedback system, consisting of youth and caregiver progress measures.
  The UP-A is an emotion-focused, transdiagnostic approach for adolescents (ages 12-18) with a primary emotional disorder. Clinicians present all skills in the context of the emotions most salient to presenting concerns and adolescent/caregiver conceptualizations of treatment needs, thereby personalizing treatment. The UP-A is delivered in 8-21 weekly sessions, with clinician flexibility regarding the sequencing and depth with which various sections are presented to clients and caregivers, as well as the emotions targeted during the course of the intervention.
Period: Overall Study
Arm/Group | Unified Protocol for Adolescents (UP-A) | Treatment as Usual Plus (TAU+) | Treatment as Usual (TAU)
Started | 68 | 60 | 68
Midpoint (8 Weeks) | 54 | 52 | 55
Post (16 Weeks) | 49 | 43 | 53
Follow-up (28 Weeks) | 45 | 45 | 52
Completed | 45 | 45 | 52
Not Completed | 23 | 15 | 16
Not completed — Withdrawal by Subject | 10 | 7 | 6
Not completed — Lost to Follow-up | 13 | 8 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Unified Protocol for Adolescents (UP-A) | Treatment as Usual Plus (TAU+) | Treatment as Usual (TAU) | Total
Number analyzed (Participants) | 68 | 60 | 68 | 196
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.69 (1.56) | 14.87 (1.76) | 14.43 (1.72) | 14.65 (1.68)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 20 | 18 | 27 | 65
  Female | 47 | 40 | 41 | 128
  Transgender (Female to Male) | 1 | 1 | 0 | 2
  Other | 0 | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 21 | 29 | 81
  Not Hispanic or Latino | 37 | 39 | 39 | 115
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 15 | 17 | 13 | 45
  White | 47 | 32 | 39 | 118
  More than one race | 2 | 8 | 9 | 19
  Unknown or Not Reported | 4 | 1 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Clinical Global Impression - Improvement (CGI-I) Scores
Description: This is a independent evaluator rated measure of improvement in symptoms and functioning. The CGI-I has a total range from 1-7 with the lower scores indicating more improvement in functioning.
Time Frame: At 16 weeks, at 28 weeks.
Population: Not all participants were able to complete the CGI-I Questionnaire at Post Visit (16 Weeks) and at Follow Up Visit (28 weeks).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unified Protocol for Adolescents (UP-A) | Treatment as Usual Plus (TAU+) | Treatment as Usual (TAU)
Number analyzed (Participants) | 46 | 41 | 49
score on a scale
  Post (16 weeks) | 2.85 (.965) | 3.20 (1.167) | 3.02 (.878)
  Follow-up (28 weeks): number analyzed (Participants) | 45 | 40 | 49
  Follow-up (28 weeks) | 2.47 (.894) | 2.45 (.904) | 2.76 (1.128)
Statistical Analysis 1: Comparison: Unified Protocol for Adolescents (UP-A) vs Treatment as Usual Plus (TAU+); DV = CGI-I at Post-Treatment; Test type: Superiority; p = .338, Mixed Models Analysis — Threshold: p < .05; Mean Difference (Net) = -.19, 95% CI 2-sided [-.58 to .20], Standard Error of Mean .20 — A negative value for the mean difference indicates that the lower numbered Group has a lower mean than the higher numbered group
Statistical Analysis 2: Comparison: Treatment as Usual Plus (TAU+) vs Treatment as Usual (TAU); DV = CGI-I at Post Treatment; Test type: Superiority; p = 0.425, Mixed Models Analysis — Threshold: p <.05; Mean Difference (Net) = 0.16, 95% CI 2-sided [-0.24 to 0.57], Standard Error of Mean .20 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Unified Protocol for Adolescents (UP-A) vs Treatment as Usual Plus (TAU+); DV = CGI-I at Post; Test type: Superiority; p = 0.09, Mixed Models Analysis — Threshold: p < .05; Mean Difference (Net) = -0.36, 95% CI 2-sided [-0.77 to 0.06], Standard Error of Mean .21 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Unified Protocol for Adolescents (UP-A) vs Treatment as Usual (TAU); DV = CGI-I at Follow-Up; Test type: Superiority; p = 0.126, Mixed Models Analysis — Threshold: p < .05; Mean Difference (Net) = -0.32, 95% CI 2-sided [-0.72 to 0.09], Standard Error of Mean 0.20 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Treatment as Usual Plus (TAU+) vs Treatment as Usual (TAU); DV = CGI-I at Follow-Up; Test type: Superiority; p = 0.28, Mixed Models Analysis — Threshold: p < .05; Mean Difference (Net) = -0.23, 95% CI 2-sided [-0.65 to 0.19], Standard Error of Mean .21 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Unified Protocol for Adolescents (UP-A) vs Treatment as Usual Plus (TAU+); DV = CGI-I at Follow-Up; Test type: Superiority; p = 0.697, Mixed Models Analysis — Threshold: p < .05; Mean Difference (Net) = -0.08, 95% CI 2-sided [-0.51 to 0.34], Standard Error of Mean .21 — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Clinical Global Impression - Severity (CGI-S) Scores
Description: This is a independent evaluator rated measure of severity of symptoms. The CGI-S has a total range from 1-7 with the higher scores indicating higher symptom severity.
Time Frame: At 16 weeks, at 28 weeks.
Population: Not all participants were able to complete the CGI-S Questionnaire at Post Visit (16 Weeks) and at Follow Up Visit (28 weeks).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unified Protocol for Adolescents (UP-A) | Treatment as Usual Plus (TAU+) | Treatment as Usual (TAU)
Number analyzed (Participants) | 46 | 41 | 49
score on a scale
  Post (16 weeks) | 4.39 (1.341) | 4.71 (1.230) | 4.41 (1.153)
  Follow-up (28 weeks): number analyzed (Participants) | 45 | 40 | 49
  Follow-up (28 weeks) | 3.98 (1.559) | 4.00 (1.396) | 4.02 (1.377)
Statistical Analysis 1: Comparison: Unified Protocol for Adolescents (UP-A) vs Treatment as Usual (TAU); DV = CGI-S at Follow-Up; Test type: Superiority; p = 0.779, Mixed Models Analysis — Threshold: p < .05; Mean Difference (Net) = -0.08, 95% CI 2-sided [-0.6 to 0.45], Standard Error of Mean .26 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Treatment as Usual Plus (TAU+) vs Treatment as Usual (TAU); DV = CGI-S at Follow-Up; Test type: Superiority; p = 0.66, Mixed Models Analysis — Threshold: p < .05; Mean Difference (Net) = 0.12, 95% CI 2-sided [-0.42 to 0.67], Standard Error of Mean .27 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Unified Protocol for Adolescents (UP-A) vs Treatment as Usual Plus (TAU+); DV = CGI-S at Post; Test type: Superiority; p = 0.629, Mixed Models Analysis — Threshold: p < .05; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.51 to 0.31], Standard Error of Mean .21 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Unified Protocol for Adolescents (UP-A) vs Treatment as Usual (TAU); DV = CGI-S at Post; Test type: Superiority; p = 0.938, Mixed Models Analysis — Threshold: p < .05; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.41 to 0.38], Standard Error of Mean .20 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Treatment as Usual Plus (TAU+) vs Treatment as Usual (TAU); DV = CGI-S at Post; Test type: Superiority; p = 0.68, Mixed Models Analysis — Threshold: p < .05; Mean Difference (Net) = 0.09, 95% CI 2-sided [-0.32 to 0.49], Standard Error of Mean .21 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Unified Protocol for Adolescents (UP-A) vs Treatment as Usual Plus (TAU+); DV = CGI-S at Follow-Up; Test type: Superiority; p = 0.479, Mixed Models Analysis — Threshold: p < .05; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.75 to 0.35], Standard Error of Mean .28 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Children's Global Assessment Scale (CGAS) Scores
Description: This is a independent evaluator rated measure of global functional impairment.The GCAS has a total range from 1-100 with the higher scores indicating better functioning.
Time Frame: At 16 weeks, at 28 weeks.
Population: Not all participants were able to complete the CGAS Questionnaire at Post Visit (16 Weeks) and at Follow Up Visit (28 weeks).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unified Protocol for Adolescents (UP-A) | Treatment as Usual Plus (TAU+) | Treatment as Usual (TAU)
Number analyzed (Participants) | 46 | 41 | 49
score on a scale
  Post (16 weeks) | 53.22 (9.575) | 52.05 (9.047) | 52.29 (8.571)
  Follow-up (28 weeks): number analyzed (Participants) | 45 | 40 | 49
  Follow-up (28 weeks) | 56.51 (12.230) | 56.76 (12.056) | 56.00 (11.281)
Statistical Analysis 1: Comparison: Unified Protocol for Adolescents (UP-A) vs Treatment as Usual (TAU); DV = CGAS at Post; Test type: Superiority; p = 0.852, Mixed Models Analysis — Threshold: p < .05; Mean Difference (Net) = 0.3, 95% CI 2-sided [-2.85 to 3.45], Standard Error of Mean 1.58 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Treatment as Usual Plus (TAU+) vs Treatment as Usual (TAU); DV = CGAS at Post; Test type: Superiority; p = 0.917, Mixed Models Analysis — Threshold: p < .05; Mean Difference (Net) = -0.17, 95% CI 2-sided [-3.41 to 3.07], Standard Error of Mean 1.62 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Unified Protocol for Adolescents (UP-A) vs Treatment as Usual Plus (TAU+); DV = CGAS at Post; Test type: Superiority; p = 0.778, Mixed Models Analysis — Threshold: p < .05; Mean Difference (Net) = 0.47, 95% CI 2-sided [-2.81 to 3.74], Standard Error of Mean 1.66 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Unified Protocol for Adolescents (UP-A) vs Treatment as Usual (TAU); DV = CGAS at Follow-Up; Test type: Superiority; p = 0.66, Mixed Models Analysis — Threshold: p < .05; Mean Difference (Net) = 0.95, 95% CI 2-sided [-3.3 to 5.19], Standard Error of Mean 2.12 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Treatment as Usual Plus (TAU+) vs Treatment as Usual (TAU); DV = CGAS at Follow-Up; Test type: Superiority; p = 0.935, Mixed Models Analysis — Threshold: p < .05; Mean Difference (Net) = -0.18, 95% CI 2-sided [-4.55 to 4.19], Standard Error of Mean 2.19 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Unified Protocol for Adolescents (UP-A) vs Treatment as Usual Plus (TAU+); DV = CGAS at Follow-Up; Test type: Superiority; p = 0.615, Mixed Models Analysis — Threshold: p < .05; Mean Difference (Net) = 1.13, 95% CI 2-sided [-3.29 to 5.55], Standard Error of Mean 2.21 — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: 28 weeks.
Arm/Group | Unified Protocol for Adolescents (UP-A) | Treatment as Usual Plus (TAU+) | Treatment as Usual (TAU)
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/60 | 0/68
Serious Adverse Events (participants affected / at risk) | 5/68 | 2/60 | 1/68
Other Adverse Events (participants affected / at risk) | 0/68 | 0/60 | 0/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Unified Protocol for Adolescents (UP-A) (N=68) | Treatment as Usual Plus (TAU+) (N=60) | Treatment as Usual (TAU) (N=68)
Hospitalization due to Suicidality (Psychiatric disorders) | 3 | 1 | 1
Suicidal behavior (Psychiatric disorders) | 2 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-13): https://cdn.clinicaltrials.gov/large-docs/66/NCT02567266/Prot_SAP_001.pdf
  • Informed Consent Form (2019-09-16): https://cdn.clinicaltrials.gov/large-docs/66/NCT02567266/ICF_000.pdf